CLINICAL TRIAL: NCT02959866
Title: Evaluating the Implementation and Impact of an Online Tool Used Within Primary Care to Improve the Income Security of Patients With Complex Health and Social Needs in Ontario and Manitoba
Brief Title: Implementation and Impact of an Online Tool Used in Primary Care to Improve Income Security
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SMH2016
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Social Determinants of Health; Poverty; Social Isolation; Social Marginalization
MeSH Terms: conditions — Social Isolation; Social Marginalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Online income tool (Experimental): Patients who complete the online income tool with their health provider during the study period.
  Interventions: Other: online income tool

INTERVENTIONS:
Other: online income tool — An online tool that uses information about the patient to develop a tailored list of financial benefits that they are eligible to apply for.
  Other Names: benefits screening tool

SUMMARY:
We will evaluate the acceptability, feasibility and impact of an online tool that helps patients identify financial benefits that they are entitled to at six clinic sites over a three month period. We will answer the following questions: Is an online tool that addresses income security feasible and acceptable to clinicians? Can such a tool be integrated into regular clinic workflow? What is the patient perspective on the tool and what is the short-term impact?

DETAILED DESCRIPTION:
Addressing the social determinants of health of patients has been identified as a key way to achieve health system goals. However, few evidence-based interventions exist. This study emerges from an ongoing collaboration between family physicians, researchers and a charitable financial literacy organization. This study aims to answer the following questions: Is an online tool that addresses income security feasible and acceptable to clinicians? Can such a tool be integrated into regular clinic workflow? What is the patient perspective on the tool and what is the short-term impact? We will recruit six primary care sites in Toronto and Winnipeg that serve low-income communities. We will introduce clinicians to screening for poverty and increasing access to additional income sources via government benefits. Following an initial orientation session, health providers will be encouraged to use the tool with any patient seen. The health provider and patient will complete the online tool together, generating a tailored list of financial benefits, along with local community resources to assist with obtaining these benefits. A brief survey on this experience will be administered to patients after they complete the tool, as well as a request to contact them in one month. Those who agree to be contacted will be interviewed on whether the intervention impacted their knowledge and ability to access benefits. We will administer an online survey to providers and conduct provider focus groups at each site at the end of study. An advisory group made up of patients living on low incomes and representatives from community agencies will support this study. An online tool could help health providers in improving the income security of their patients. Strengths of this study include that it involves a diverse set of clinics and that the tool has been implemented pragmatically, in the real world of busy primary care clinics. Limitations include the convenience sampling method, that the selected clinics may not be representative of all primary care providers and the relatively short follow-up period. Our findings will provide insight into the potential of electronic tools that assist providers address the social determinants of health.

ELIGIBILITY:
Inclusion Criteria:

* Used the online income tool with their health provider
* Able to provide consent
* Able to converse in English
* Able to be reached by telephone or email

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Pinto, MD MSc, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - Department of Family Medicine, Faculty of Medicine, University of Manitoba, Winnipeg, Manitoba
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Background] Aery A, Rucchetto A, Singer A, Halas G, Bloch G, Goel R, Raza D, Upshur REG, Bellaire J, Katz A, Pinto AD. Implementation and impact of an online tool used in primary care to improve access to financial benefits for patients: a study protocol. BMJ Open. 2017 Oct 22;7(10):e015947. doi: 10.1136/bmjopen-2017-015947. PMID 29061603

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Clinicians will be encouraged to screen patients for poverty and use the online tool with every eligible patient during 3-months. It is difficult to estimate how many patients will be seen during the 3-month time period, the number who will be living in poverty, the number who agree to the intervention and be consented to the study for follow-up.
Groups:
- Online Income Tool: Patients who complete the online income tool with their health provider during the study period and were enrolled in the study through participation in the evaluation.
  Online income tool: An online tool that uses information about the patient to develop a tailored list of financial benefits that they are eligible to apply for.
Period: Overall Study
Arm/Group | Online Income Tool
Started | 59
Telephone Interview at 1 Month Follow-up | 59
Completed | 58
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: This is the sample of people who were enrolled in this research by participating in one-month follow-up interviews after using the tool with their healthcare provider.
Groups:
- Online Income Tool: Patients who were reached for follow-up at one month, after using the Online income tool with their healthcare provider: 59
  online income tool: An online tool that uses information about the patient to develop a tailored list of financial benefits that they are eligible to apply for.
Arm/Group | Online Income Tool
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants] — Population: We did not collect information about age during our follow-up interviews with participants.
Sex: Female, Male [Count of Participants; unit: Participants] — We did not collect data on sex. Population: We did not collect information on gender from those reached for follow-up interviews.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 59
Region of Enrollment [Number; unit: participants]
  Canada | 59
Whether participants have trouble making ends meet at the end of the month [Count of Participants; unit: Participants] | 59

OUTCOME MEASURES:

1. Primary Outcome: Awareness of Financial Benefits
Description: Self-reported awareness of at least one financial benefit
Time Frame: 4 weeks
Population: This the the number of people who used the tool to completion with their healthcare provider
Measure: Count of Participants; unit: Participants
Groups:
- Online Income Tool: Patients who finished using the tool with their healthcare providers and produced a PDF of recommended benefits that they may have been eligible to apply for.
  online income tool: An online tool that uses information about the patient to develop a tailored list of financial benefits that they are eligible to apply for.
Arm/Group | Online Income Tool
Number analyzed (Participants) | 59
Participants | 59

2. Secondary Outcome: Increase in Income
Description: Self-reported increase in income through accessing a financial benefit
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Online Income Tool: Patients who complete the online income tool with their health provider during the study period and were reached for an interview at 1 month follow-up.
  Online income tool: An online tool that uses information about the patient to develop a tailored list of financial benefits that they are eligible to apply for.
Arm/Group | Online Income Tool
Number analyzed (Participants) | 59
Participants | 10

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Online Income Tool
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT02959866/Prot_SAP_000.pdf